CLINICAL TRIAL: NCT01482403
Title: A Phase II, Randomized, Double-Blind, Multicenter, Parallel Group Study to Evaluate the Sustained Virologic Response of the HCV Polymerase Inhibitor Prodrug RO5024048 in Combination With Boceprevir and Pegasys®/Copegus® in Patients With Chronic Hepatitis C Genotype 1 Virus Infection Who Were Prior Null Responders to Treatment With Pegylated Interferon/Ribavirin
Brief Title: A Study of Mericitabine in Combination With Boceprevir and Pegasys/Copegus in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV27780; 2011-002714-37 (EudraCT Number)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; 2'-fluoro-2'-methyl-3',5'-diisobutyryldeoxycytidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Treatment Arm A (Experimental): 24 weeks of therapy with mericitabine 1000 mg twice a day (BID), boceprevir 800 mg three times daily (TID), Pegasys 180 microgram/week, and Copegus 1000/1200 mg/day (total treatment duration of 24 weeks), followed by a 24-week treatment-free follow-up period.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: boceprevir; Drug: mericitabine
- Treatment Arm B (Experimental): 24 weeks of therapy with mericitabine + boceprevir + Pegasys/Copegus followed by 24 weeks of therapy with boceprevir + Pegasys/Copegus (triple) (total treatment duration of 48 weeks), followed by a 24-week treatment-free follow-up period.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: boceprevir; Drug: mericitabine
- Treatment Arm C (Control) (Active Comparator): 4 weeks of therapy with mericitabine placebo, boceprevir placebo + Pegasys/Copegus, then 20 weeks of therapy with mericitabine placebo + boceprevir + Pegasys/Copegus, then 24 weeks of therapy with boceprevir + Pegasys/Copegus (total treatment duration of 48 weeks), followed by a 24-week treatment-free follow-up period.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: mericitabine placebo; Drug: boceprevir placebo; Drug: boceprevir

INTERVENTIONS:
Drug: Copegus — total daily dose of 1000 mg or 1200 mg for 24 weeks
  Arms: Treatment Arm A
Drug: Copegus — total daily dose of 1000 mg or 1200 mg for 48 weeks
  Arms: Treatment Arm B; Treatment Arm C (Control)
Drug: Pegasys — 180 microgram subcutaneous once a week for 24 weeks
  Arms: Treatment Arm A
Drug: Pegasys — 180 microgram subcutaneous once a week for 48 weeks
  Arms: Treatment Arm B; Treatment Arm C (Control)
Drug: boceprevir — 800 mg three times a day for 24 weeks
  Arms: Treatment Arm A
Drug: boceprevir — 800 mg three times a day for 48 weeks
  Arms: Treatment Arm B
Drug: mericitabine — 1000 mg twice daily for 24 weeks
  Arms: Treatment Arm A; Treatment Arm B
Drug: mericitabine placebo — mericitabine placebo
  Arms: Treatment Arm C (Control)
Drug: boceprevir placebo — boceprevir placebo
  Arms: Treatment Arm C (Control)
Drug: boceprevir — 800 mg three times a day for 44 weeks
  Arms: Treatment Arm C (Control)

SUMMARY:
This randomized, double-blind, multi-center, placebo-controlled, parallel-group study will evaluate the sustained virologic response and the safety of mericitabine (RO5024048) in combination with boceprevir and Pegasys/Copegus in patients with chronic hepatitis C infection. The anticipated time on study treatment is up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Chronic hepatitis C infection for at least 6 months duration
* Hepatitis C genotype 1a or 1b
* Patients must have discontinued prior hepatitis C treatment at least 12 weeks prior to enrollment in this study
* Patient showed a previous null response to therapy as defined by < 2 log10 IU/mL decrease in viral titer after at least 12 weeks of treatment with PEG-IFN/RBV

Exclusion Criteria:

* Hepatitis C infection with a genotype other than genotype 1a or 1b
* Body mass index <18 or >/=36
* Hepatitis A, hepatitis B, or HIV infection
* Herbal remedies </=1 month prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response 12 weeks after treatment (SVR-12) | up to 60 weeks

SECONDARY OUTCOMES:
Sustained virological response 4 weeks after treatment | up to 52 weeks
Virologic response over time | 60 weeks
Proportion of patients who develop treatment resistance | 60 weeks
Safety (incidence of adverse events) | 60 weeks
Pharmacokinetics: trough concentration of RO4995855 | Day 1 and Week 8
Pharmacokinetics: trough concentration of RO5012433 | Day 1 and Week 8
Pharmacokinetics: trough concentration of boceprevir | Day 1 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- United States (7):
  - Littleton, Colorado
  - Chicago, Illinois
  - Shreveport, Louisiana
  - Detroit, Michigan
  - Kansas City, Missouri
  - San Antonio, Texas
  - Chesapeake, Virginia
- Canada (3):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - London, Ontario
- France (3):
  - Créteil
  - Nice
  - Rennes
- Germany (3):
  - Berlin
  - Hamburg
  - Hanover
- Italy (3):
  - Napoli, Campania
  - Milan, Lombardy
  - Florence, Tuscany
- Ponce, Puerto Rico
- Spain (4):
  - Palma de Mallorca, Balearic Islands
  - Santander, Cantabria
  - Pontevedra, Pontevedra
  - Valencia, Valencia

REFERENCES:
- [Derived] Wedemeyer H, Forns X, Hezode C, Lee SS, Scalori A, Voulgari A, Le Pogam S, Najera I, Thommes JA. Mericitabine and Either Boceprevir or Telaprevir in Combination with Peginterferon Alfa-2a plus Ribavirin for Patients with Chronic Hepatitis C Genotype 1 Infection and Prior Null Response: The Randomized DYNAMO 1 and DYNAMO 2 Studies. PLoS One. 2016 Jan 11;11(1):e0145409. doi: 10.1371/journal.pone.0145409. eCollection 2016. PMID 26752189